CLINICAL TRIAL: NCT00270803
Title: The Effects of Marijuana on Orientation and Motor Coordination and Brain Metabolism in Regular Smokers of Marijuana.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Dr. Michal Roll, Sourasky Medical Center Tel Aviv
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: TASMC-05-EE-03-124-CTIL
Record Dates: First submitted 2005-12-25; First posted 2005-12-28 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2005-12

CONDITIONS: Marijuana Dependence
Keywords: Marijuana, FDG, PET, maze, THC, motor coordination.
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Placebo Comparator): Low nicotine cigarettes without THC
  Interventions: Drug: Tetra Hydro Cannabinol (THC)

INTERVENTIONS:
Drug: Tetra Hydro Cannabinol (THC) — Oral THC 13mg and 17mg smoked in low nicotine cigarettes
  Other Names: Marijuana, cannabis

SUMMARY:
This study investigates the effects of 17mg and 13mg Delta THC on orientation and motor coordination and brain metabolic activity in regular users of marijuana. Subjects were tested twice, after smoking cigarettes with marijuana and after smoking cigarettes without marijuana.On both occasions they performed on a virtual reality maze task. They were afterwards scanned in Positron Emission Tomography (PET) with Fluoro-deoxy-glucose (FDG).

DETAILED DESCRIPTION:
This study investigates the effects of 17mg and 13mg Delta THC on orientation and motor coordination and brain metabolic activity in regular users of marijuana. Subjects were tested twice, after smoking cigarettes with marijuana and after smoking cigarettes without marijuana. On both occasions they performed on a virtual reality maze task. They were afterwards scanned in Positron Emission Tomography (PET) with Fluoro-deoxy-glucose (FDG). 12 subjects were tested so far on both conditions.

ELIGIBILITY:
Inclusion Criteria:

* Marijuana dependence
* Age 20-65
* Male and female

Exclusion Criteria:

* Pregnant women
* Dependence on other substances
* Psychiatric diagnosis apart from marijuana dependence
* Neurological disorder
* Young persons

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Brain metabolic activity (FDG) | 30-40 minutes

SECONDARY OUTCOMES:
Reaction time (RTs) and errors in performance | 40 minutes
Subjective ratings on visual analog scale | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Aviv M Weinstein, Ph.D, Principal Investigator — Sourasky Medical Center; Einat Even-Sapir, M.D. Ph.D, Principal Investigator — Sourasky Medical Center
Locations (1):
- Department of Nuclear Medicine, Tel Aviv, Israel